CLINICAL TRIAL: NCT04184258
Title: Treatment of Systemic Lupus Erythematosus With Pooled Allogenic Olfactory Mucosa Derived Mesenchymal Stem Cells
Brief Title: Treatment of Systemic Lupus Erythematosus With Pooled Allogenic Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSC1(SLE)
Record Dates: First submitted 2019-12-01; First posted 2019-12-03 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; mesenchymal stem cells
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLE patients MSC treatment (Experimental): Patients with SLE, who receive pooled mesenchymal stem cells in addition to the standard treatment according to the Clinical protocols
  Interventions: Biological: Pooled mesenchymal stem cell; Other: Standard treatment according to the Clinical protocols
- SLE patients standard treatment (Active Comparator): Patients with SLE, who receive standard treatment according to the Clinical protocols
  Interventions: Other: Standard treatment according to the Clinical protocols

INTERVENTIONS:
Biological: Pooled mesenchymal stem cell — Pooled allogenic mesenchymal stem cell derived from olfactory mucosa
  Arms: SLE patients MSC treatment
Other: Standard treatment according to the Clinical protocols — Standard SLE treatment according to the Clinical protocols approved by the Ministry of healthcare of Republic of Belarus

SUMMARY:
Treatment of systemic lupus erythematosus with pooled allogenic mesenchymal stem cells

ELIGIBILITY:
Inclusion Criteria:

* SLE diagnosis (4 of 11 criteria by ACR);
* positive dsDNA;
* SELENA-SLEDAI index ≥6;
* active lupus nephritis;
* patient can read, understand and follow the procedures.

Exclusion Criteria:

* need for dialysis;
* planned renal transplantation;
* any medical condition which can be associated with the high risk for the patient;
* pregnancy/lactation;
* chronic infections, including hepatitis B/C, tuberculosis, HIV;
* any malignant tumor in the last 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluation | 6 month
  Efficacy evaluation (SELENA-SLEDAI)

SECONDARY OUTCOMES:
Safety eveluation | 1 month
  Absence of adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, Dr, Study Director — Director, the Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus; Konstantin A Chizh, Dr, Study Director — Associate professor, Belarusian State Medical University
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus